CLINICAL TRIAL: NCT05920551
Title: Efficacy of Gastrocnemius Stretching on Plantar Heel Pain, Foot Mobility and Function in Patients With Plantar Fasciitis: A Randomised Controlled Trial
Brief Title: Gastrocnemius Stretching on Plantar Heel Pain, Foot Mobility and Function in Patients With Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/7080002023
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Plantar Fascitis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastrocnemius Stretching Group (Experimental): Patients will receive ultrasound therapy, fascia strengthening exercises, and gastrocnemius stretching exercises.
  Interventions: Other: Gastrocnemius Stretching Exercises; Other: Standard care
- Control Group (Active Comparator): Patients will receive ultrasound therapy and fascia strengthening exercises without gastrocnemius stretching exercises.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Gastrocnemius Stretching Exercises — The gastrocnemius stretching exercises will be performed by patients in the study group. These exercises will involve stretching the gastrocnemius muscle in a controlled manner to improve flexibility and reduce tension in the plantar fascia.
  Arms: Gastrocnemius Stretching Group
Other: Standard care — Ultrasound therapy: A therapeutic ultrasound device will be used to apply ultrasound waves to the plantar fascia area for pain relief and to promote healing. The frequency, intensity, and duration of the ultrasound therapy will be determined by the treating physical therapist based on individual patient needs.Fascia strengthening exercises: Patients will be instructed to perform exercises targeting the intrinsic foot muscles and the plantar fascia to improve strength and function. Examples of these exercises include toe curls, towel scrunches, and arch lifts. Patients will be asked to perform these exercises daily, with the specific number of repetitions and sets determined by the physical therapist.

SUMMARY:
The study aims to investigate the effectiveness of gastrocnemius stretching exercises on plantar heel pain intensity, foot mobility, and function in patients with plantar fasciitis.

DETAILED DESCRIPTION:
This randomized controlled trial will include patients diagnosed with plantar fasciitis. Participants will be randomly assigned to either a study group performing gastrocnemius stretches or a control group. Both groups will receive ultrasound therapy and fascia strengthening exercises. The study group will additionally perform specific gastrocnemius stretching exercises. Outcome measures will be assessed before and after 4 weeks of intervention and will include pain intensity, foot mobility using an inversion/eversion device, and function using the Foot and Ankle Ability Measure. The study hypothesizes that the study group will demonstrate greater improvements in pain, foot mobility, and function compared to the control group. The study findings could guide physical therapy interventions for patients with plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

1. Pain reproduced with palpation of the plantar fascia
2. localized and sharp but not radiating
3. worse in the initial step after and an extended period of rest
4. decreased initially after the first steps but exacerbated with increased activityat least 6 weeks
5. unresponsive conservative form of plantar fasciitis care (ie, rest, stretching, full-length silicone insole, prescription NSAIDs when taken for a period of 2 weeks)

Exclusion Criteria:

1. history of previous steroid injections
2. previous surgery of the foot, lumbar spine disc herniation or back injury
3. patients with rheumatic diseases (e.g., rheumatoid arthritis, spondyloarthropathy, gout disease, enthesopathy, Sjogren's syndrome, and systemic lupus erythematosus)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Plantar heel pain intensity | Changes in Plantar heel pain intensity at Baseline and after 4 weeks of intervention and 3 months
  Measured using a Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Changes in Foot mobility | Changes in foot mobility at Baseline and after 4 weeks of intervention and 3 months
  Measured using an inversion/eversion device
Changes in Foot function | Changes in foot function at Baseline and after 4 weeks of intervention and 3 months
  Measured using the Foot and Ankle Ability Measure (FAAM)

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No